CLINICAL TRIAL: NCT03371693
Title: A Phase III Clinical Trail of Cytoreductive Surgery(CRS) Plus Hyperthermic Intraperitoneal Chemotherapy(HIPEC) With Lobaplatin in Advanced and Recurrent Epithelial Ovarian Cancer
Brief Title: Cytoreductive Surgery(CRS) Plus Hyperthermic Intraperitoneal Chemotherapy(HIPEC) With Lobaplatin in Advanced and Recurrent Epithelial Ovarian Cancer
Acronym: HIPECOV
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, CAI Hongbing, Professor of Wuhan University, MD, PhD, Chef of the Department of Gynecological Oncology of Zhongnan Hospital, member of the standing committee of Chinese Gynecologic Cancer Society, Zhongnan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIPECOV
Record Dates: First submitted 2017-11-27; First posted 2017-12-13 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Ovarian Cancer; Ovary Neoplasm; Ovarian Neoplasms; Epithelial Ovarian Cancer; Ovarian Cancer, Epithelial; Hyperthermic Intraperitoneal Chemotherapy(HIPEC)
Keywords: hyperthermic intraperitoneal chemotherapy; epithelial ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIPEC (Experimental): Patients will undergo a CRS plus HIPEC and IVCT. Hyperthermic intraperitoneal chemotherapy (HIPEC) is a procedure in which the abdominal cavity is bathed in a warm solution of anti-cancer medications for 60 minutes.
  A single drug lobaplatin(30mg/m2)will be administered in normal saline via HIPEC and it will be continued for 60 minutes in the hyperthermic phase (41°C-43°C). HIPEC will be performed at the 1st, 3rd and 5th day after CRS. The intravenous chemotherapy(IVCT) will start from 7th-14th day after CRS.
  Interventions: Device: HIPEC; Device: CRS; Device: IVCT
- Non HIPEC (Other): Patients will undergo only CRS and IVCT. Patients will receive standard platinum-based combination doublet chemotherapy for 6-8 cycles after CRS.
  Interventions: Device: CRS; Device: IVCT

INTERVENTIONS:
Device: HIPEC — Patients consenting to this protocol will undergo their scheduled surgical procedure. After cytoreductive surgery (CRS) to a residual disease ≤ 2.5 mm, a single dose of lobaplatin (30 mg/m2) will be administered in normal saline via intraperitoneal hyperthermic perfusion using the closed-abdomen technique. HIPEC will be continued for 60 minutes in the hyperthermic phase (43℃±0.5℃). And HIPEC will be repeated at the 3 and 5 day after the day of CRS plus HIPEC.
  Arms: HIPEC
Device: CRS — cytoreductive surgery (CRS) to a residual disease ≤ 2.5 mm.
Device: IVCT — platinum-based intravenous chemotherapy

SUMMARY:
A phase III prospective study with the primary objective to compare the efficacy and safety of HIPEC( Hyperthermic Intraperitoneal Chemotherapy). The target population for this study is patients with primary or recurrence ovarian, peritoneal or fallopian tube cancers undergoing CRS( Cytoreductive Surgery). Patients will be divided into two groups. Group A will undergo CRS plus HIPEC and then go on to receive standard platinum-based combination doublet intravenous chemotherapy. Group B will undergo CRS and then go on to intravenous chemotherapy.

DETAILED DESCRIPTION:
This is a phase III prospective study with the primary objective to compare the efficacy and safety of HIPEC. The target population for this study is patients with primary or recurrence ovarian, peritoneal or fallopian tube cancers undergoing CRS. 'Platinum-sensitive' recurrence is defined as recurrence 6 months after the completion of the primary platinum-based chemotherapy. A single dose of lobaplatin 40mg/m2 will be administered via HIPEC , and will be administered at the time of surgery, 3 days after surgery and 5 days after surgery. Patients of group A will undergo CRS plus HIPEC and then go on to receive standard platinum-based combination doublet intravenous chemotherapy (carboplatin and paclitaxel, carboplatin and gemcitabine, or carboplatin and liposomal doxorubicin) for 6 cycles. Patients of group B will undergo CRS and then go on to intravenous chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75
* Karnofsky performance status >50 or World Health Organization performance score < 2
* primary or recurrence ovarian, peritoneal or fallopian tube epithelial cancer; first intra-abdominal recurrence without distant metastasis (including: unique resectable pleural metastasis which are platinum-sensitive; resectable single lymphatic metastasis retroperitoneal or inguinal)
* preoperative platinum-based chemotherapy (carboplatin and paclitaxel, carboplatin and liposomal doxorubicin, gemcitabine, trabectedin or topotecan)
* lesion can be removed completely or residual disease < 0.5 cm
* last chemotherapy finished no more than 12 weeks after surgery
* no hepatic function damage
* white blood cell count ≥3.5*10^9/L; platelet count ≥80*10^9/L; Hemoglobin ≥90g/L
* no contraindication of surgery and anesthesia
* life expectancy ≥ 3 months

Exclusion Criteria:

* age < 18 or >75
* no history of other cancer
* platinum allergy
* distant metastasis
* used anti-angiogenic drug within 8 weeks
* possibility of more than two resection of alimentary canal
* recurrence < 6 months after primary treatment
* histologic type: non epithelial origin
* infection out of control
* follow-up unable to carry on (geographic or psychic)
* cardiac insufficiency or respiratory insufficiency
* has received HIPEC already
* being in other clinical study
* pregnancy or lactation period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival rate | 5 years
  assess overall survival rate in 5 years in both arms
1 year survival rate | 1 year
  assess the survival rate in 1 year for both arms
3 year survival rate | 3 years
  assess the survival rate in 3 years for both arms

SECONDARY OUTCOMES:
Progression-free survival | 5 years
  assess the Progression-free survival rate during 5 years for both study arms
quality of life | 5 years after CRS or until death
  Patients will fill the EORTC Quality of life questionaire-C30 form to measure the quality of life after a standard treatment.
postoperative complication | 5 years
  measured with physical examination and/or computed tomography（CT）and/or ultrasound examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China